CLINICAL TRIAL: NCT07045324
Title: A Comparative Study on the Effect of Vagus Nerve Stimulation and Ischemic Compression on Trapezius Trigger Points
Brief Title: Effect of Vagus Nerve Stimulation on Trapezius Trigger Point
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Shahla Hassanilar Ansaroudi, Principal Investigator,Mcs. Physiotherapy and Rehabilitation Department ,Bahçeşehir University, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAU-MA25
Record Dates: First submitted 2025-06-04; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Myofascial Pain Syndrome; Trigger Points
Keywords: Trigger points; Vagus Nerve Stimulation; Parasympathetic System
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Vagus Nerve Stimulation; Acupressure; Exercise

STUDY DESIGN:
Intervention Model Description: This study employs a parallel assignment model with three distinct intervention arms. Ninety participants with trigger points in the upper trapezius muscle are randomly assigned to one of three groups (n=30 each): non-invasive vagus nerve stimulation (nVNS), ischemic compression (trigger point massage), or exercise (control). Each group receives their respective intervention over 10 sessions (3 times per week for 4 weeks). The parallel design ensures that participants remain in their assigned group throughout the study, with no crossover. Outcomes, including pain intensity, trigger point number, pain pressure threshold, neck function, well-being, and functional mobility, are assessed at baseline and post-intervention (week 4). Single blinding (outcomes assessor) is implemented to minimize bias in outcome measurements.
Who Masked: Outcomes Assessor
Masking Description: This study employs single blinding, where the outcomes assessors are masked to the participants' group assignments. Participants are randomized into one of three groups (non-invasive vagus nerve stimulation, ischemic compression, or exercise), and the interventions are administered by unblinded study personnel. To minimize bias, assessors responsible for measuring outcomes, including pain intensity (Visual Analog Scale), number of trigger points, pain pressure threshold (algometer), neck function (Copenhagen Neck Functional Disability Scale), well-being (WHO-5 Well-Being Index), and functional mobility, are unaware of the intervention each participant receives. Participants and intervention providers are not blinded due to the nature of the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Vagus Nerve Stimulation (nVNS) (Experimental): Participants receive non-invasive auricular vagus nerve stimulation bilaterally to the concha and tragus using a TENS-based device (10 Hz, 300 µs, 20 minutes per session) for 10 sessions over 4 weeks, with intensity adjusted to patient comfort.
  Interventions: Device: Vagus Nerve Stimulation (nVNS)
- Arm 2: Ischemic Compression (Active Comparator): Participants receive manual trigger point massage (ischemic compression) applied to trapezius trigger points for 30-90 seconds per point, 3 times per week for 10 sessions.
  Interventions: Procedure: Ischemic Compression
- Exercise (Control) (Active Comparator): Participants perform a standardized exercise program including isometric neck exercises, upper trapezius stretching, and chin tuck exercises, conducted 3 times per week for 10 sessions.
  Interventions: Behavioral: Exercise (Control)

INTERVENTIONS:
Device: Vagus Nerve Stimulation (nVNS) — Arm 1 (Vagus Nerve Stimulation (nVNS)) is an experimental intervention, as it tests a novel approach (non-invasive vagus nerve stimulation) for trigger point treatment.
  Arms: Arm 1: Vagus Nerve Stimulation (nVNS)
Procedure: Ischemic Compression — Arm 2 (Ischemic Compression) is an active comparator, as it uses a standard treatment (trigger point massage) commonly applied for myofascial pain.
  Arms: Arm 2: Ischemic Compression
Behavioral: Exercise (Control) — Arm 3 (Exercise (Control)) is explicitly labeled as the control group in your document, using a standard exercise program, which aligns with an active comparator (since it's an active intervention rather than a placebo or no intervention).
  Arms: Exercise (Control)

SUMMARY:
This randomized controlled trial aimed to evaluate the efficacy of non-invasive vagus nerve stimulation (nVNS) compared to ischemic compression (trigger point massage) and exercise in treating trigger points in the upper trapezius muscle. Ninety participants aged 18-55 with at least two trigger points were randomly assigned to three groups: nVNS, ischemic compression, or exercise (control). Interventions were administered over 10 sessions (3 times per week). Outcomes included pain intensity (Visual Analog Scale, VAS), trigger point number, pain pressure threshold (algometer), neck function (Copenhagen Neck Functional Disability Scale, KBFÖS), well-being (WHO-5 Well-Being Index), and functional mobility. The nVNS group demonstrated statistically significant improvements in all outcomes compared to the other groups (p < 0.05).

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is characterized by trigger points-hyperirritable spots in skeletal muscle associated with pain, stiffness, and reduced function. The upper trapezius muscle is a common site for trigger points, contributing to neck pain and disability. Traditional treatments include ischemic compression and exercise, but non-invasive vagus nerve stimulation (nVNS) has emerged as a promising modality due to its ability to modulate pain pathways and autonomic function.

This study investigated whether nVNS is more effective than ischemic compression or exercise in reducing pain and improving function in patients with trapezius trigger points. Participants were randomized into three groups (n=30 each)

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years.
* Presence of at least two trigger points (active or latent) in the upper trapezius muscle, confirmed by palpation.
* Ability to provide informed consent.

Exclusion Criteria:

* History of cervical spine surgery or trauma.
* Neurological disorders (e.g., epilepsy, stroke).
* Pregnancy or breastfeeding.
* Use of pacemakers or other implanted electrical devices.
* Active infection or skin lesions at the stimulation site.
* Recent use of botulinum toxin or other trigger point injections.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (VAS)(Visual Analog Scale ) | Baseline and post-intervention (week 4)
  Measured using the Visual Analog Scale (0-10 ), where 0 indicates no pain and 10 indicates worst possible pain.
Number of Trigger points | Measurements were taken pre- and post-intervention.(week 4)
  Count of active and latent trigger points in the upper trapezius muscle, assessed by palpation.
Pain Pressure Threshold (Algometer) | Measurements were taken pre- and post-intervention. (week 4)
  Measured using a digital algometer (kg/cm²) at trigger point sites to assess pain sensitivity.
Neck Function (CNFDS(Copenhagen Neck Functional Disability) | Measurements were taken pre- and post-intervention. (week 4)
  Assessed using the Copenhagen Neck Functional Disability Scale, evaluating neck-related disability (0-30, higher scores indicate greater disability).
WHO-5(World Health Organization-Five Well-Bing Index) | Measurements were taken pre- and post-intervention. (week 4)
  Description: Measured using the WHO-5 Well-Being Index, a 5-item scale (0-25, higher scores indicate better well-being)

CONTACTS AND LOCATIONS:
Overall Officials: Hasankerem Alptekin, Prof.DR, Study Director — Bahçeşehir University
Locations (1):
- Bahçeşehir University, Physiotherapy and Rehabilitation, Istanbul, Helthy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
"No individual participant data (IPD) will be shared due to privacy and ethical considerations, in accordance with institutional policies."

REFERENCES:
- [Result] Xu A, Huang Q, Rong J, Wu X, Deng M, Ji L. Effectiveness of ischemic compression on myofascial trigger points in relieving neck pain: A systematic review and meta-analysis. J Back Musculoskelet Rehabil. 2023;36(4):783-798. doi: 10.3233/BMR-220045. PMID 36872769
- [Result] Moraska AF, Schmiege SJ, Mann JD, Butryn N, Krutsch JP. Responsiveness of Myofascial Trigger Points to Single and Multiple Trigger Point Release Massages: A Randomized, Placebo Controlled Trial. Am J Phys Med Rehabil. 2017 Sep;96(9):639-645. doi: 10.1097/PHM.0000000000000728. PMID 28248690
- [Result] Alghadir AH, Iqbal A, Anwer S, Iqbal ZA, Ahmed H. Efficacy of Combination Therapies on Neck Pain and Muscle Tenderness in Male Patients with Upper Trapezius Active Myofascial Trigger Points. Biomed Res Int. 2020 Mar 10;2020:9361405. doi: 10.1155/2020/9361405. eCollection 2020. PMID 32258159

DOCUMENTS (1):
  • Study Protocol (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT07045324/Prot_000.pdf